CLINICAL TRIAL: NCT01754675
Title: Cardiovascular Effects of a Soccer Match in Viewers With With Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Cardiologia de Santa Catarina (Other)
Responsible Party: Principal Investigator, Daniel Medeiros Moreira, MD. MSc., Instituto de Cardiologia de Santa Catarina
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 03807212.5.0000.0113
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soccer (Experimental): Watching the soccer match at the time that the favorite team is playing
  Interventions: Behavioral: Soccer
- Movie (Placebo Comparator): Watching a movie at the time that the favorite team is playing
  Interventions: Behavioral: Movie

INTERVENTIONS:
Behavioral: Soccer — Watching the soccer match at the time that the favorite team is playing
  Arms: Soccer
Behavioral: Movie — Watching a movie at the time that the favorite team is playing
  Arms: Movie

SUMMARY:
Watching football matches could cause increased blood pressure and heart rate induced by catecholamines and thus increase the incidence of cardiovascular events. However, no studies have evaluated the responses of blood pressure and heart rate in soccer spectators.

This study evaluates the hemodynamic response in Brazilian soccer fans suffering from coronary artery disease during a dispute over a game of your favorite team.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease;
* Avai or Figueirense (brazilian soccer teams) fans

Exclusion Criteria:

* Acute coronary syndrome in less than 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Average mean arterial pressure | 90 minutes
  To evaluate the difference between the average mean arterial pressure in patients with coronary artery disease, or not watching a game of soccer your favorite team;

SECONDARY OUTCOMES:
Mean heart rate | 90 minutes
  To evaluate the difference between the mean heart rate;
Systolic blood pressure | 90 minutes
  To evaluate the difference between the systolic blood pressure;
Diastolic blood pressure | 90 minutes
  To evaluate the difference between the diastolic blood pressure;
Double product | 90 minutes
  To evaluate the difference between the double product (the product of heart rate and systolic blood pressure);
Angina | 90 minutes
  To evaluate the difference between the presence of angina;

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Moreira, MD. MSc., Study Chair — Instituto de Cardiologia de Santa Catarina
Locations (1):
- Instituto de Cardiologia de Santa Catarina, São José, Santa Catarina, Brazil